CLINICAL TRIAL: NCT02204072
Title: A Phase Ib/II, Multicentre, Open Label, Randomized Study of BI 836845 in Combination With Enzalutamide, Versus Enzalutamide Alone, in Metastatic Castration-Resistant Prostate Cancer (CRPC) Following Disease Progression on Docetaxel-Based Chemotherapy and Abiraterone
Brief Title: BI836845 Plus Enzalutamide in Castrate Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1280.8; 2013-004011-41 (EudraCT Number)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — xentuzumab; enzalutamide

ARMS (2):
- BI 836845 & Enzalutamide (Experimental)
  Interventions: Drug: BI 836845; Drug: Enzalutamide
- Enzalutamide (Active Comparator)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: BI 836845
  Arms: BI 836845 & Enzalutamide
Drug: Enzalutamide
  Arms: Enzalutamide
Drug: Enzalutamide
  Arms: BI 836845 & Enzalutamide

SUMMARY:
The overall aim of the trial is to investigate the safety and anti-tumour activity of an experimental drug BI 836845 taken together with the prostate cancer drug, enzalutamide, compared to enzalutamide given alone, in castrate resistant prostate cancer (CRPC) patients that have previously been treated and failed on docetaxel and abiraterone treatments. Initially, a tolerability and safety phase (phase Ib escalation) will be performed to confirm the maximum tolerated dose (MTD), or recommended doses of both BI 836845 and enzalutamide that can be taken together.

Once the MTD, or recommended phase II dose, have been determined an expansion cohort will also be explored (phase Ib expansion) in CRPC patients already taking enzalutamide and have a rise in prostate serum antigen (PSA) levels. Patients may not have received prior docetaxel or abiraterone. Patients in this cohort will receive the MTD, or recommended phase II dose, of BI 836845 and enzalutamide determined in the phase Ib escalation phase.

The randomised trial (phase II) will be an open label, parallel group study design in a 1:1 ratio to which patients will receive either BI 836845 plus enzalutamide (Arm A) at the MTD/recommended doses, or enzalutamide alone (Arm B).

In all parts of the trial safety, anti-tumour activity will be assessed, in addition to circulating tumour cells (CTC), prostate serum antigen (PSA) response and progression, and determination of Overall Survival (OS).

ELIGIBILITY:
Inclusion criteria:

* The patient has histologically, or cytologically, confirmed adenocarcinoma of the prostate.
* Male patient aged, equal to, or more than,18 years old.
* Patients with radiographic evidence of metastatic prostate cancer (stage M1 or D2). Distant metastases evaluable by radionuclide bone scan, CT scan, or MRI within 28 days before the start of study treatment.
* Patients with a prostate serum antigen (PSA), equal to, or more than, 5 nanograms per mililiter (ng/mL).
* Patients with prior surgical or chemical castration with a serum testosterone of <50 ng/mL. If the method of castration is luteinizing hormone releasing level hormone (LHRH) agonists, the patient must be willing to continue the use of LHRH agonists during protocol treatment.
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* Cardiac left ventricular function with resting ejection fraction >50% as determined by echocardiogram (ECHO) or multigated acquisition scan (MUGA).
* Absolute neutrophil count (ANC) >=1500/microlitre (uL).
* Haemoglobin >=9 gram per deciliter (g/dL).
* Platelets >=100,000/uL.
* Bilirubin <= 1.5 times the upper limit of normal (ULN).
* Aspartate transaminase (AST) and alanine transaminase (ALT) <= 2.5 times the ULN(or <= 5 times the ULN if liver metastases are present).
* Creatinine <= 1.5 x ULN.
* International normalized ratio (INR) </= 2 and a partial thromboplastin time (PTT) </= 5 seconds above the ULN (unless on oral anticoagulant therapy). Patients receiving full dose anticoagulation therapy are eligible provided they meet all other criteria, are on a stable dose of oral anticoagulant or low molecular weight heparin (except warfarin or coumarin-like anticoagulants, which are not permitted).
* Fasting plasma glucose < 8.9 millimols per liter (mmol/L) (< 160 milligrams per deciliter (mg/dL) and glycated haemoglobin (hemoglobin A1c (HbA1c)) < 8.0%.

Inclusion criteria only for patients entering phase Ib escalation and phase II:

* Patients who have disease progression during, or after, receiving docetaxel and have had at least 12 weeks of treatment and in the opinion of the investigator are unlikely to derive significant benefit from additional docetaxel-based therapy, or were intolerant to therapy with this agent.
* Patients who have disease progression during, or after, receiving abiraterone treatment in any setting.
* Patients must have progressive disease defined as at least one of the following:

  1. Progressive measurable disease: using conventional solid tumour criteria RECIST 1.1.
  2. Bone scan progression: at least two new lesions on bone scan, plus a rising PSA as described in (c) below.
  3. Increasing PSA level: at least two consecutive rising PSA values over a reference value (PSA #1) taken at least 1 week apart. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2.

Inclusion criterion only for patients entering phase Ib expansion cohort:

* Patients must be receiving continuous enzalutamide treatment and show a rise in PSA level: at least two consecutive rising PSA values over a reference value (PSA #1) taken at least 1 week apart. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2.
* Archive tumour tissue is available prior to recruitment for pharmacogenomic tests

Exclusion criteria:

* Prior therapy with agents targeting Insulin Growth Factor (IGF) and/or Insulin Growth Factor Receptor (IGFR) pathway.
* Patients that have been treated with any of the following within 4 weeks of starting trial treatment: chemotherapy, immunotherapy, biological therapies, molecular targeted, hormone therapy (except LHRH agonists and LHRH antagonists), radiotherapy (except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within 2 weeks prior to study treatment).
* Use of any investigational drug within 4 weeks before start of trial treatment or concomitantly with this trial.
* Patients that have been treated with strong cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8) inhibitors, CYP2C8 inducers, within 2 weeks of starting the trial treatment.
* Fridericia´s Corrected QT interval (QTcF) prolongation > 450 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome). The QTcF will be calculated as the mean of the 3 ECGs taken at screening.
* Patients with small cell or neuroendocrine tumours.
* Patients with known or suspected leptomeningeal metastases.
* Uncontrolled or poorly controlled hypertension.
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness.
* Patients with epilepsy, seizures, or predisposing factors for seizure as judged by the investigator.
* Patients unable to comply with the protocol as judged by the investigator.
* Active alcohol or active drug abuse as judged by the investigator.
* A history of allergy to human monoclonal antibodies.
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception, e.g. condom plus spermicide use for participating males, plus another form of birth control such as implants, injectables, combined oral contraceptives, intrauterine devices for female partners, during the trial and for at least three months after end of active therapy. Men unwilling to agree to not donate sperm while on trial drug and up to 6 months following the last dose of trial drug.
* Previous or concomitant malignancies at any other site with the exception of the following:

  * benign basal cell carcinoma
  * benign low grade transitional cell carcinoma of the bladder
  * other effectively treated malignancy that has been in remission for more than 5 years and is considered to be cured
* Only for patients entering phase Ib dose escalation and phase II cohorts:
* Patients who have received more than 2 prior non-docetaxel containing cytotoxic chemotherapy regimens for Metastatic Castration-Resistant Prostate Cancer (mCRPC).
* Patients who have received a taxane based treatment or abiraterone, within 4 weeks before start of study treatment.
* Patients that have received prior enzalutamide in any setting will not be eligible.

Exclusion criterion only for patients entering phase Ib expansion cohort:

- Patients that have received prior taxane-based chemotherapy or abiraterone in any setting will not be eligible for the expansion cohort.

Additional exclusion criterion for patients undergoing tumour biopsy:

* For patients that are to undergo the tumour biopsy, a history of a hereditary bleeding disorder, or clinically relevant major bleeding event in the past 6 months, as judged by the investigator.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- United States (3):
  - Karmanos Cancer Institute, Detroit, Michigan
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Oregon Health and Sciences University, Portland, Oregon
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Netherlands (2):
  - Erasmus MC - Daniel den Hoed, Rotterdam
  - Tweesteden Ziekenhuis, locatie Tilburg, Tilburg
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - OncoCare Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Instituto Valenciano de Oncología, Valencia
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - The Clatterbridge Cancer Centre, Bebington, Wirral
  - Velindre Cancer Centre, Cardiff
  - The Christie Hospital, Manchester
  - Churchill Hospital, Oxford
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicentre, open-label, randomised study to determine the safety, tolerability and anti-tumour activity of xentuzumab (BI 836845) in combination with enzalutamide in patients with advanced prostate cancer that has spread. The trial consists of 3 parts: Phase 1b dose escalation part, Phase 1b expansion part, Phase 2 two arm, parallel design.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated
Groups:
- Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide: 750 milligram (mg) xentuzumab (10mg/milliliter (mL)) was supplied in 20mL vials and diluted in physiological sodium chloride solution (0.9%)) as liquid formulation was administered as weekly 1-hour intravenous (i.v.) infusion on Days 1, 8, 15 and 22 together with four liquid-filled soft gelatin capsules of 40mg (total: 160mg) enzalutamide administered orally once daily during each 28-day cycle of treatment until disease progression or occurrence of undue toxicities. Infusion duration of xentuzumab could be extended to more than 1 hour in case of infusion reaction or adverse events. Phase Ib escalation part.
- Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide: 1000 milligram (mg) xentuzumab (10mg/mL was supplied in 20mL vials and diluted in physiological sodium chloride solution (0.9%)) as liquid formulation was administered as weekly 1-hour intravenous (i.v.) infusion on Days 1, 8, 15 and 22 together with four liquid-filled soft gelatin capsules of 40mg (total: 160mg) enzalutamide administered orally once daily during each 28-day cycle of treatment until disease progression or occurrence of undue toxicities. Infusion duration of xentuzumab could be extended to more than 1 hour in case of infusion reaction or adverse events. Phase Ib escalation part.
- Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide: 1000 milligram (mg) xentuzumab (10mg/mL was supplied in 20mL vials and diluted in physiological sodium chloride solution (0.9%)) as liquid formulation was administered as weekly 1-hour intravenous (i.v.) infusion on Days 1, 8, 15 and 22 together with four liquid-filled soft gelatin capsules of 40mg (total: 160mg) enzalutamide administered orally once daily during each 28-day cycle of treatment until disease progression or occurrence of undue toxicities. Infusion duration of xentuzumab could be extended to more than 1 hour in case of infusion reaction or adverse events. Phase Ib expansion part.
- Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide: 1000 milligram (mg) xentuzumab (10mg/mL was supplied in 20mL vials and diluted in physiological sodium chloride solution (0.9%)) as liquid formulation was administered as weekly 1-hour intravenous (i.v.) infusion on Days 1, 8, 15 and 22 together with four liquid-filled soft gelatin capsules of 40mg (total: 160mg) enzalutamide administered orally once daily during each 28-day cycle of treatment until disease progression or occurrence of undue toxicities. Infusion duration of xentuzumab could be extended to more than 1 hour in case of infusion reaction or adverse events. Phase II part.
- Phase II: 160 mg Enzalutamide: Four liquid-filled soft gelatin capsules of 40mg (total: 160mg) enzalutamide administered orally once daily during each 28-day cycle of treatment until disease progression or occurrence of undue toxicities. Phase II part.
Period: Overall Study
Arm/Group | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Started | 3 | 7 | 24 | 43 | 43
Treated | 3 | 7 | 24 | 43 | 43
Discontinued Xentuzumab Due to Progressive Disease | 2 | 4 | 21 | 24 | 0
Discontinued Xentuzumab Due to Adverse Event | 0 | 3 | 0 | 7 | 0
Discontinued Xentuzumab Due to Withdrawal by Subject | 1 | 0 | 2 | 9 | 0
Discontinued Xentuzumab Due to Other Reason | 0 | 0 | 1 | 1 | 0
Completed (Completed=Number of patients on treatment) | 0 (Number of patients on Xentuzumab+Enzalutamide) | 0 (Number of patients on Xentuzumab+Enzalutamide) | 0 (Number of patients on Xentuzumab+Enzalutamide) | 2 (Number of patients on Xentuzumab+Enzalutamide) | 0 (Number of patients on Enzalutamide)
Not Completed | 3 | 7 | 24 | 41 | 43
Not completed — Discontinued Enzalutamide due to withdrawal by subject | 1 | 0 | 2 | 9 | 6
Not completed — Discontinued Enzalutamide due to adverse events | 0 | 3 | 1 | 6 | 6
Not completed — Discontinued Enzalutamide due to progressive disease | 2 | 4 | 19 | 26 | 31
Not completed — Discontinued Enzalutamide due to other reason | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide | Total
Number analyzed (Participants) | 3 | 7 | 24 | 43 | 43 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.67 (11.85) | 70.71 (7.09) | 73.38 (7.81) | 68.58 (8.80) | 69.91 (7.92) | 70.14 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 7 | 24 | 43 | 43 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 5 | 12 | 21
  Not Hispanic or Latino | 3 | 7 | 20 | 37 | 31 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 7 | 23 | 27 | 33 | 93
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Prostate Surface Antigen (PSA) at baseline [Mean (Standard Deviation); unit: Micorgram / Liter] — Population: Phase 1b escalation part and Phase 1b expansion part: Treated Set. Phase II: Randomised Set.
  Micorgram / Liter
    number analyzed (Participants) | 3 | 7 | 24 | 43 | 42 | 119
    (all) | 272.03 (100.38) | 437.99 (390.02) | 113.59 (252.65) | 671.23 (935.44) | 562.97 (1592.71) | 496.77 (1120.62)

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib Escalation Part: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: Number of patients with DLTs were used to determine the maximum tolerated dose (MTD) in the Phase Ib escalation part. The MTD in this study was defined as the highest protocol dose level of xentuzumab in combination with enzalutamide, at which no more than 1 out of 6 patients in a cohort experienced a DLT during the MTD evaluation period.
Time Frame: From first administration of xentuzumab up to start of Cycle 2, up to 28 days.
Population: MTD-set: The MTD set defined the set of patients in the Phase Ib escalation part who were fully evaluable for determination of the MTD in the first treatment course. 1 patient in the 1000 mg Xentuzumab + 160 mg Enzalutamide arm was not evaluable for the MTD determination due to missed doses. Phase Ib escalation part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Phase Ib Escalation Part: Maximum Tolerated Dose (MTD) Based on the Occurrence of Dose Limiting Toxicity (DLT) During the First Treatment Course
Description: Maximum tolerated dose (MTD) based on the occurrence of dose limiting toxicity (DLT) during the first treatment course. The MTD in this study was defined as the highest protocol dose level of xentuzumab in combination with enzalutamide, at which no more than 1 out of 6 patients in a cohort experienced a DLT during the MTD evaluation period.
Time Frame: From first administration of xentuzumab up to start of Cycle 2, up to 28 days.
Population: as for outcome 1
Measure: Number; unit: Milligram
Groups:
- Xentuzumab + Enzalutamide: This arm comprises all dose groups from Phase Ib escalation phase (750 mg Xentuzumab + 160 mg Enzalutamide and 1000 mg Xentuzumab + 160 mg Enzalutamide)
Arm/Group | Xentuzumab + Enzalutamide
Number analyzed (Participants) | 9
Milligram | 1000

3. Primary Outcome: Phase Ib Expansion Part: Prostate Specific Antigen (PSA) Response
Description: The primary endpoint of the Phase Ib expansion part was PSA response. PSA response was defined as a decline in PSA value >50% compared to baseline which was confirmed by the next available value occurring at least 3 weeks later. The confirmatory value had to be at least 50% lower than the baseline, but could be higher than the first PSA value taken into account for response. However the confirmatory value was not allowed to be 50% higher than this first PSA value. If it was ≥ 50% higher than the first PSA value, the next available sample was to be taken to determine if response had been achieved. The date of response was the date that the first 50% (or greater) decline was observed. Number of participants with response is reported.
Time Frame: At Cycle 1 Day 1 before study treatment and from Cycle 3 Day 1 and Day 1 of every cycle thereafter until the end of treatment, up to 35 months.
Population: Treated Set (TS): All patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1). Phase Ib expansion part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide
Number analyzed (Participants) | 24
Participants
  Yes, Confirmed | 1
  Yes, Unconfirmed | 1
  No | 21
  Missing | 1

4. Primary Outcome: Phase II Part: Progression Free Survival (PFS) Based on Investigator Assessment
Description: PFS was defined as the time from randomisation until radiological tumour progression in bone (based on Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria) or soft tissue (based on modified RECIST 1.1) or death from any cause, whichever occurred earlier. Clinical disease progression was not considered for determination of a PFS event, unless the outcome of the progression was death. Median PFS time in months is reported.
  PFS was calculated as follows:
  For patients with 'event' as an outcome for PFS (according to modified RECIST version 1.1 or PCWG2):
  PFS [days] = date of outcome - date of randomisation + 1.
  For patients with 'censored' as an outcome for PFS (according to modified RECIST version 1.1 or PCWG2):
  PFS (censored) [days] = date of outcome - date of randomisation + 1.
Time Frame: From randomisation until radiological tumor progression or death from any cause, whichever occurred earlier, up to 1269 days.
Population: Randomised Set (RS): All randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Phase II part.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Months | 7.4 [3.5 to 8.7] | 6.2 [3.5 to 11.1]
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.9549, Two-sided log-rank test; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.57 to 1.70] — Cox proportional hazard model. Hazard ratio: Comparison vs Enzalutamide

5. Secondary Outcome: Phase Ib Expansion Part: Progression Free Survival (PFS) Based on Investigator Assessment
Description: PFS was defined as the time from randomisation until radiological tumour progression in bone (based on Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria) or soft tissue (based on modified RECIST 1.1) or death from any cause, whichever occurred earlier. Clinical disease progression was not considered for determination of a PFS event, unless the outcome of the progression was death. Median PFS time in months is reported.
  PFS was calculated as follows:
  For patients with 'event' as an outcome for PFS: (according to modified RECIST version 1.1 or PCWG2) PFS [days] = date of outcome - date of first treatment administration + 1.
  For patients with 'censored' as an outcome for PFS (according to modified RECIST version 1.1 or PCWG2):
  PFS (censored) [days] = date of outcome - date of first treatment administration + 1.
Time Frame: From first treatment administration of any study medication until radiological tumor progression or death from any cause, whichever occurred earlier, up to 1114 days.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide
Number analyzed (Participants) | 24
Months | 8.2 [3.5 to 14.6]

6. Secondary Outcome: Phase Ib Expansion Part: Changes in Circulating Tumour Cells (CTC) Response - CTC Reduction From >=5 to <5 Cells Per 7.5 mL Blood for at Least One Post-baseline Time Point
Description: Changes in circulating tumour cells (CTC) response - CTC reduction from >=5 to <5 cells per 7.5 mL blood for at least one post-baseline time point. Number of participants with CTC Response (yes/no) is reported.
Time Frame: Prior to study drug administration at Day 1 Cycle 1, Day 1 Cycle 2, Day 1 Cycle 3, Day 1 Cycle 5, Day 1 Cycle 7 and every 12 weeks thereafter, up to end of treatment. Up to 35 months.
Population: Treated Set (TS): All patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1). Only participants with baseline CTC value >= 5 cells per 7.5mL were included in the analysis. Phase Ib expansion part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide
Number analyzed (Participants) | 9
Participants
  Yes | 1
  No | 8

7. Secondary Outcome: Phase II Part: Radiological Progression Free Survival (PFS), Based on Central Review
Description: as for outcome 5
Time Frame: as for outcome 4
Population: Randomised Set: All randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Phase II part.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Months | 3.6 [3.5 to 8.1] | 7.1 [3.6 to 8.2]
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.5425, Two-sided log-rank test; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.68 to 2.06] — Cox proportional hazards model. Hazard ratio: Comparison vs. Enzaludamide

8. Secondary Outcome: Phase II Part: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from randomisation to death from any cause. Median survival time in months is reported.
  Overall survival at cut-off date for final analysis (24-Oct-2019) is reported.
Time Frame: From randomisation until radiological tumor progression or death from any cause (until cut-off date for final analysis), whichever occurred earlier, up to 1269 days.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Months | 13.6 [8.7 to 19.4] | 13.6 [8.7 to 21.3]
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.5534, Two-sided log-rank test; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.71 to 1.90] — Cox proportional hazards model. Hazard ratio: Comparison vs. Enzalutamide

9. Secondary Outcome: Phase II Part: Time to Prostate Specific Antigen (PSA) Progression
Description: For the definition of time to PSA progression, the following rules are used:
  * Decline from baseline in PSA before increasing: Time to PSA progression is defined as the time from the date of randomisation until the date where a 25% or greater increase in PSA and an absolute increase of 2 ng/mL or more from baseline, is documented (which is confirmed by the next available value occurring at least 3 weeks later).
  * No decline from baseline in PSA: Time to PSA progression is defined as the time from the date of randomisation until the date where a 25% or greater increase in PSA and an absolute increase of 2 ng/mL or more from baseline, is documented. However, only values after 12 weeks of therapy are considered.
  Time to PSA progression [days] = date of PSA progression - date of randomisation + 1.
  For patients not presenting with PSA progression or being lost to follow-up:
  Time to PSA progression (censored) [days] = date of censoring - date of randomisation + 1.
Time Frame: At screening, at Cycle 1 Day 1 and from Cycle 3 Day 1 and at Day 1 of every cycle thereafter until end of treatment, up to 40.1 months.
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Months | 4.6 [2.8 to 5.7] | 3.7 [2.8 to 4.6]
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.1514, Two-sided log-rank test; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.35 to 1.18] — Cox proportional hazards model. Hazard ratio: Comparison vs. Enzalutamide

10. Secondary Outcome: Phase II Part: Maximum Decline in Prostate Specific Antigen (PSA)
Description: Maximum decline in (PSA) compared to baseline. The maximum decline in PSA is defined as the change in PSA between the baseline PSA value and the minimum post-baseline PSA value. The change from baseline is defined as: Change from baseline in PSA (ng/mL) = PSA value post-baseline - PSA value at baseline.
  Maximum decline in PSA is defined as:
  Maximum decline in PSA (ng/mL) = min(PSA value post-baseline) - PSA value at baseline.
Time Frame: as for outcome 9
Population: Randomised Set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Only participants with non-missing values were included in the analysis. Phase II part.
Measure: Mean (Standard Deviation); unit: Microgram / Liter
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 40 | 37
Microgram / Liter | -102.20 (580.59) | -94.13 (1020.31)

11. Secondary Outcome: Phase II Part: Percentage Change in Prostate Specific Antigen (PSA) at Week 12
Description: Percentage change in PSA from baseline to Week 12. Percentage change in PSA from baseline to week 12 of treatment is defined as:
  Percentage change in PSA (%) = 100*(PSA value at week 12 - PSA value at baseline)/PSA value at baseline
  For this assessment, it is allowed to take a value:
  * until one week later than week 12, in case the PSA assessment was delayed
  * one day earlier due to the one day window allowed by the protocol Values from assessments between day 84 and day 92 after first treatment administration will therefore be taken into account (according to the protocol schedule for visits at week 12).
Time Frame: At baseline and at Week 12.
Population: Randomised Set: All randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Only participants with non-missing values were included in the analysis. Phase II part.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 31 | 30
Percentage change | 10.13 (83.25) | 49.72 (109.91)

12. Secondary Outcome: Phase II Part: Prostate Specific Antigen (PSA) Response
Description: PSA response - defined as a decline in PSA value >50% (which is confirmed by a second value 3 to 4 weeks apart).
  PSA response was defined as a decline in PSA value >50% compared to baseline which was confirmed by the next available value occurring at least 3 weeks later. The confirmatory value had to be at least 50% lower than the baseline, but could be higher than the first PSA value taken into account for response. However the confirmatory value was not allowed to be 50% higher than this first PSA value. If it was ≥ 50% higher than the first PSA value, the next available sample was to be taken to determine if response had been achieved. Number of participants with response is reported.
Time Frame: At Cycle 1 Day 1 and from Cycle 3 Day 1 and at Day 1 of every cycle thereafter until end of treatment, up to 40.1 months.
Population: Randomised Set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Phase II part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Participants
  Yes - confirmed | 7 | 8
  Yes - unconfirmed | 2 | 0
  No | 31 | 29
  Missing | 3 | 6

13. Secondary Outcome: Phase II Part: Circulating Tumour Cells (CTC) Reduction Defined as CTC Decline From ≥5 to <5 Cells Per 7.5 mL Blood for at Least One Post-baseline Time-point
Description: CTC reduction is defined as CTC decline from ≥5 to <5 cells per 7.5 mL blood for at least one post-baseline time-point. Patients with a CTC value < 5 cells per 7.5mL blood at baseline, or with missing baseline values were not taken into consideration for this endpoint. Baseline value is the value collected before a patient starts treatment with trial medication.
  Number of participants per category is reported.
Time Frame: Prior to study drug administration at Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 5 Day 1, Cycle 7 Day 1 and then every 12 weeks thereafter, until end of treatment. Up to 40.1 months.
Population: Randomised Set (RS): This patient set included all randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Only patients with baseline CTC value >=5 cells per 7.5mL were included in the analysis. Phase II part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 25 | 19
Participants
  Yes | 4 | 2
  No | 19 | 15
  Missing on treatment | 2 | 2
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.6186, Regression, Logistic; Odds ratio, p-value and confidence interval were obtained from logistic regression model; Odds Ratio (OR) = 1.579, 95% CI 2-sided [0.269 to 12.515]

14. Secondary Outcome: Phase II Part: Maximum Decline (%) in Circulating Tumour Cells (CTC) Counts
Description: Maximum decline in CTC counts (in number of cells) compared with baseline that occurred at any point after treatment start , defined as the difference between the minimum post-baseline CTC value and the baseline CTC value. Patients with missing baseline value are considered missing for this criterion. Baseline value is the value collected before a patient starts treatment with trial medication. Positive values for maximum decline in CTC are possible in case no decline in CTC occurred. This indicates an increase in CTC.
Time Frame: as for outcome 13
Population: Randomised Set: All randomised patients in the Phase II part, regardless of whether or not they received treatment. Patients were assigned to xentuzumab in combination with enzalutamide or enzalutamide alone. Only participants with baseline CTC value were included in the analysis. Phase II part.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 32 | 28
Percentage (%) | 41.96 (289.085) | 21.33 (201.353)

15. Secondary Outcome: Phase II Part: Circulating Tumour Cells (CTC) Status at Week 12
Description: CTC status (≥5 or <5 cells per 7.5mL blood) at Week 12. Number of participants per category is reported.
Time Frame: At Week 12.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
Number analyzed (Participants) | 43 | 43
Participants
  ≥5 cells per 7.5ml blood | 26 | 20
  <5 cells per 7.5ml blood | 11 | 16
  Missing on treatment | 6 | 7
Statistical Analysis 1: Comparison: Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide vs Phase II: 160 mg Enzalutamide; Test type: Other; p = 0.1920, Regression, Logistic; Odds Ratio (OR) = 1.891, 95% CI 2-sided [0.727 to 5.059] — Odds ratio, p-value and confidence interval were obtained from logistic regression model

ADVERSE EVENTS:
Time Frame: [All cause mortality]: Up to 430 days for Phase 1b escalation, up to 1107 days Phase 1b expansion and up to 1322 days for Phase II part. [Serious and other Adverse events]. From first drug administration until last drug administration + residual effect period of 42 days, up to 370 days for Phase 1b escalation, up to 1107 days for Phase 1b expansion, up to 1262 days for Phase II.
Description: Treated Set (TS): This patient set included all patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (from Day 1).
  All-cause mortality includes all death throughout the whole study period, also including death reports after the cut-off date of the final analysis.
Arm/Group | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide | Phase II: 160 mg Enzalutamide
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/7 | 0/24 | 34/43 | 31/43
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/7 | 8/24 | 19/43 | 17/43
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 24/24 | 43/43 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide (N=3) | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=7) | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=24) | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=43) | Phase II: 160 mg Enzalutamide (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Condition aggravated (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 2 | 2 | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Escalation: 750 mg Xentuzumab + 160 mg Enzalutamide (N=3) | Phase Ib Escalation: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=7) | Phase Ib Expansion: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=24) | Phase II: 1000 mg Xentuzumab + 160 mg Enzalutamide (N=43) | Phase II: 160 mg Enzalutamide (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 15 | 19
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 5 | 5 | 11 | 14
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 10 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 8 | 11 | 12
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 9 | 9
Asthenia (General disorders) | 0 | 0 | 3 | 7 | 11
Fatigue (General disorders) | 3 | 5 | 9 | 29 | 21
Oedema peripheral (General disorders) | 0 | 1 | 3 | 2 | 4
Pain (General disorders) | 0 | 1 | 0 | 3 | 6
Peripheral swelling (General disorders) | 0 | 0 | 3 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 4 | 5
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 4 | 5
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 6 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 4 | 3 | 5
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 3 | 3 | 2
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 | 3
Weight decreased (Investigations) | 2 | 2 | 4 | 16 | 5
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 9 | 26 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 14 | 13 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 12 | 13 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 2 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 5 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 7 | 10
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 5 | 5 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 3 | 3
Headache (Nervous system disorders) | 0 | 1 | 6 | 3 | 4
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 4 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 4
Somnolence (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 1 | 0 | 1 | 3
Depressed mood (Psychiatric disorders) | 0 | 1 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 3 | 2 | 6 | 7
Nightmare (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 3 | 3
Haematuria (Renal and urinary disorders) | 1 | 1 | 2 | 6 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 3
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 6 | 6
Hot flush (Vascular disorders) | 0 | 0 | 1 | 3 | 7
Hypertension (Vascular disorders) | 0 | 0 | 2 | 3 | 4
Hypotension (Vascular disorders) | 0 | 1 | 2 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 2 | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 2 | 2
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Distractibility (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT02204072/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02204072/SAP_001.pdf